CLINICAL TRIAL: NCT02054611
Title: Randomized Educational ARDS Diagnosis Study (READS)
Brief Title: The Educational ARDS Diagnosis Study
Acronym: READS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Unity Health Toronto (Other); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Eddy Fan, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: READS1
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: ARDS
Keywords: ARDS; Chest radiographs; Vignettes; Online educational video

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational Module First (Active Comparator): Respondents will complete the online educational module first, followed by the evaluation
  Interventions: Other: Online Educational Module
- Evaluation First (Placebo Comparator): Respondents will complete the the evaluation first, followed by the online educational module
  Interventions: Other: Evaluation First (Placebo)

INTERVENTIONS:
Other: Online Educational Module — A descriptive video detailing the diagnosis of ARDS according to the Berlin Definition, along with online educational materials available for review.
  Arms: Educational Module First
Other: Evaluation First (Placebo) — The respondents will view the descriptive video detailing the diagnosis of ARDS according to the Berlin Definition, along with online educational materials available for review only after they have completed the evaluation.
  Arms: Evaluation First

SUMMARY:
Without rigorous, high-quality training materials, the results of the LUNG-SAFE study examining the global incidence and outcomes of severe lung failure (acute respiratory distress syndrome [ARDS]) could be confused by either under-recognition of patients with, or misclassification of patients without, ARDS. This problem has been previously identified with the use of the prior ARDS definitions, particularly in patients with milder severity of illness. Importantly, the chest x-ray criteria in the ARDS definition has demonstrated only moderate reliability when applied by experts, although this can be improved through the use of training radiographs (as will be used in this educational module). The investigators hypothesize that the training from the educational module will allow more accurate diagnosis of ARDS by data collectors/study coordinators participating in the LUNG-SAFE study.

DETAILED DESCRIPTION:
In this LUNG-SAFE sub-study, the investigators will evaluate the effect of a brief online educational module on correctly identifying patients (i.e., standardized cases) with ARDS according to the Berlin Definition.

The investigators hypothesize that the training from the educational module will allow more accurate diagnosis of ARDS according to the Berlin Definition by participating data collectors/study coordinators.

Data collectors and study coordinators from ICUs participating in LUNG-SAFE would be randomized (by simple random number generator) to one of the following online educational streams:

1. Educational module completion followed by evaluation
2. Evaluation followed by educational module completion

Limited demographic data will be collected from the respondents, along with their responses to the 15 multiple choice test questions. Time spent viewing the educational module will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Study coordinators/data collectors for the LUNG-SAFE study

Exclusion Criteria:

* No informed consent to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
ARDS Diagnosis | up to 4 weeks
  The number of correct responses to the evaluation component (15 multiple choice questions) of the educational module (in aggregate).

SECONDARY OUTCOMES:
ARDS Diagnosis | up to 4 weeks
  Number of correct responses to the evaluation component of the educational modules, separated by question type (vignettes vs. chest x-rays)
Time | up to 4 weeks
  Amount of time spent completing the educational module

CONTACTS AND LOCATIONS:
Overall Officials: Eddy Fan, MD, PhD, Principal Investigator — University Health Network and Mount Sinai Hospital; Gordon Rubenfeld, MD, MSc, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario